CLINICAL TRIAL: NCT05759143
Title: Enhancing Information Management for Young Adults After Genetic Cancer Risk Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Nest Genomics (Industry)
Responsible Party: Principal Investigator, Jennifer Mack, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-657
Record Dates: First submitted 2023-02-24; First posted 2023-03-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Genetic Predisposition to Disease; Genetic Predisposition
Keywords: Genetic Predisposition to Disease; Genetic Predisposition; Genetic Testing; Cancer Risk Syndromes; VUS; Variant of Uncertain Significance; Pathogenic Variant
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nest Refinement Phase (Experimental): 20 participants and clinicians will complete study procedures as outlined:
  * Nest portal orientation and access.
  * Semi-structured, 30-minute interviews. Solicited feedback on content and processes will refine the intervention for a pilot phase.
  Interventions: Behavioral: Nest Platform
- Nest Pilot Phase (Experimental): 10 Participants and 10 clinicians will complete study procedures as outlined:
  * Baseline survey (participant).
  * Standard clinic visit.
  * Nest portal orientation and access (participant and clinician).
  * Post-visit survey (participant and clinician).
  * Brief, 30-minute, semi-structured interview (participant and clinician).
  Interventions: Behavioral: Nest Platform

INTERVENTIONS:
Behavioral: Nest Platform — Patient- and clinician-facing portal via secure link

SUMMARY:
This research is being done to develop the electronic platform Nest for young adults (ages 18-39) who have had prior cancer genetic testing. The platform will give patients and their clinicians access to continuously updated information about both pathogenic variants and variants of uncertain significance (VUS).

The name of the intervention used in this research study is:

Nest portal (electronic platform for patients and clinicians)

DETAILED DESCRIPTION:
The goal of the electronic platform Nest is to help patients understand and manage genetic test results and recommended care and to help clinicians with access to results and recommendations, facilitating orders, and documentation. The portal has two parts, one for participants and one for clinicians.

For the first phase of the study, participants will give their feedback on the Nest portal's content and processes that will guide refinement of the portal. The Pilot phase will test the feasibility and acceptability of the intervention.

The research study procedures include a baseline survey, using the portal after receiving a brief orientation from the study team, a follow-up survey, and then a 30-minute interview.

Participants will be in this research study for up to 2 hours.

It is expected that about 40 people will take part in this research study.

The electronic platform is being developed by Nest Genomics.

ELIGIBILITY:
Inclusion Criteria AIM 1:

* YA Patients:

  * Ages 18-39 years, inclusive.
  * Has had previous cancer genetic testing, with a finding of a pathogenic variant or VUS; patient has previously received results from the clinical team.
  * English-speaking and -reading.
  * Receiving care at DFCI.
  * Not undergoing active cancer therapy at the time of approach.
* Clinicians:

  * Cancer risk physicians (oncologists, gastroenterologists, geneticists), oncologists, nurse practitioners, physician assistants, or genetic counselors.
  * English-speaking and -reading.
  * Cares for YAs aged 18-39 with cancer risk syndromes.

Inclusion Criteria AIM 2:

* YA Patients:

  * Ages 18-39 years, inclusive.
  * Has had previous cancer genetic testing, with a finding of a pathogenic variant or VUS; patient has previously received results from the clinical team.
  * English-speaking and -reading.
  * Receiving care at Dana-Farber Cancer Institute.
  * Did not participate in a stakeholder interview (Aim 1).
  * Not undergoing active cancer therapy at the time of approach.
* Clinicians:

  * Oncologists, nurse practitioners, cancer risk physicians, or genetic counselors.
  * English-speaking and -reading.
  * Caring for a participating YA.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participant Utilization (Feasibility) | 2 hours
  Defined as > 70% of consenting participants who use the intervention.
Proportion of Clinician Utilization (Feasibility) | 2 hours
  Defined as > 70% of consenting clinicians who use the intervention.
Proportion of Clinicians with FIM (Feasibility of Intervention Measure) Score > 4 | At post-visit survey, up to 2 hours
  Defined as >70% of clinicians consider the intervention feasible as assessed by the post-visit survey.
Proportion of Participants with AIM (Acceptability of Intervention Measure) Score > 4 | At post-visit survey, up to 30 days
  Defined as > 70% of young adult participants consider the intervention successful as measured by a post-visit AIM score >4
Proportion of Clinicians with AIM Score > 4 | at post-visit survey, up to 2 hours
  Defined as > 70% of clinicians consider the intervention successful as measured by a post-visit AIM score >4

SECONDARY OUTCOMES:
Change in knowledge of cancer risk | Baseline and post visit up to 2 hours
  Change in cancer knowledge will be assessed by participant survey at baseline and post visit.
Change in Recommended screening | Baseline and post visit up to 2 hours
  Change in Recommended screening will be assessed by participant survey at baseline and post visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mack, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu